CLINICAL TRIAL: NCT00097825
Title: Efficacy and Safety of Zoledronic Acid for the Treatment of Osteoporosis in Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446M2308
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Osteoporosis
Keywords: Male Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
The goal of this study is to determine the effectiveness and safety of an annual intravenous treatment of zoledronic acid for the treatment of osteoporosis in men. All patients will receive calcium and vitamin D supplements.

ELIGIBILITY:
Inclusion Criteria:

* Male, 25-85 years old

Exclusion Criteria:

* Current users of bisphosphonates such as Aredia® (pamidronate), Didronel® (etidronate), Fosamax® (alendronate), Actonel ® (residronate), Skelid® (tiludronate)
* History of severe liver, kidney or eye disease

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 25 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288
Dates: Start 2004-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To compare % change in Lumbar Spine BMD from Baseline to Month 24 in ZOL (annual i.v. infusion) vs Alendronate (weekly oral) osteoporotic male populations

SECONDARY OUTCOMES:
To compare % change in Lumbar Spine BMD from Baseline to Months 6 and 12 in ZOL (annual i.v. infusion) vs Alendronate (weekly oral) osteoporotic male populations
To compare % change in BMD at the Total Hip, Femoral Neck, Trochanter and Total Body, from Baseline to Months 6, 12 and 24 in ZOL (annual i.v. infusion) vs Alendronate (weekly oral) osteoporotic male populations
To compare Biomarkers of bone turnover in the annual Zol i.v. and weekly alendronate populations at all study timepoints, relative to Baseline

CONTACTS AND LOCATIONS:
Locations (26):
- United States (16):
  - Catalina Pointe Clinical Research Inc., Tucson, Arizona
  - Diablo Clinical Research, Walnut Creek, California
  - Colorado Center for Bone Research, Lakewood, Colorado
  - Radiant Research, Stuart, Florida
  - United Osteoporosis Center, Gainesville, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Mercy Arthritis and Osteoporosis Center, Des Moines, Iowa
  - St. Joseph Hospital, Bangor, Maine
  - Osteoporosis and Clinical Trials Center, Hagerstown, Maryland
  - New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - Helen Hayes Hospital, West Haverstraw, New York
  - UC Bone Health and Osteoporosis Center, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Radiant Research, Wyomissing, Pennsylvania
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
- Australia (3):
  - Garvan Institute of Medical Research, Sydney, New South Wales
  - Repatriation General Hospital, Daw Park, South Australia
  - Keogh Institute for Medical Research, Nedlands, Western Australia
- Canada (7):
  - Clinical Research Center, Vancouver, British Columbia
  - QEII HealthSciences Center, Halifax, Nova Scotia
  - Charlton Medical Building, Hamilton, Ontario
  - Centre De Recherche Clinique De Laval, Laval, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Groupe de Recherche en Rhumatologie et Maladies Osseuses, Sainte-Foy, Quebec
  - Saskatoon Osteoporosis Center, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Grbic JT, Black DM, Lyles KW, Reid DM, Orwoll E, McClung M, Bucci-Rechtweg C, Su G. The incidence of osteonecrosis of the jaw in patients receiving 5 milligrams of zoledronic acid: data from the health outcomes and reduced incidence with zoledronic acid once yearly clinical trials program. J Am Dent Assoc. 2010 Nov;141(11):1365-70. doi: 10.14219/jada.archive.2010.0082. PMID 21037195
- See also: For information regarding US facilities, click this hyperlink. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?t=i&trialID=291&diseaseID=33